CLINICAL TRIAL: NCT04719728
Title: Assessment of Audiological Outcome of Cochlear Implant Program at Sohag University Hospital
Brief Title: Evaluate Audiological Outcome of Cochlear Implant Program in Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shahenda Abdelmateen Moussa, Assessment of audiological outcome of Cochlear Implant program at Sohag University Hospital, Sohag University
Other Study IDs: Soh-Med-21-01-06
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Hearing Loss, Sensorineural, Bilateral
MeSH Terms: conditions — Hearing Loss | interventions — Noise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pre lingual: aided response, speech perception threshold impedance telemetry electrically evoked action potential p1n1 cortical evoked potential
  Interventions: Diagnostic Test: Aided pure tone audiometry
- post lingual: aided response, speech perception threshold speech in noise impedance telemetry electrically evoked action potential p1n1 cortical evoked potential
  Interventions: Diagnostic Test: Aided pure tone audiometry

INTERVENTIONS:
Diagnostic Test: Aided pure tone audiometry — aided response, speech, evoked potential
  Other Names: Speech perception test; Speech in noise; P1N1 cortical evoked potential; Impedance telemetry; Electrically evoked Action Potential ECAP

SUMMARY:
Evaluation of the outcome of cochlear implantation (CI) is very important issue since adequate hearing is linked to improved communication outcomes and school performance, development of speech and language, enhances speech perception in quiet and noise and even allows CI recipients to use the telephone.

As well as there is a growing need for a widely used set of international quality standards on minimal outcome measurements to determine outcomes in CI recipients, monitor the auditory progress of CI recipients over time and to be able to relate on important issues as the most ideal age for implantation and the cut-off audiological thresholds for CI indication.

This study will be conducted to evaluate outcome of cochlear implantation in sohag university hospital.

Aim of work:

To evaluate the outcome of cochlear implantation in Sohag university hospital.

DETAILED DESCRIPTION:
Materials and Methods:

- It is a prospective study on cochlear implant recipients in sohag cochlear implant unite from 2014: 2020.

• Subjects: Cochlear implant recipients in sohag cochlear implant unite from 2014: 2020.

Subjects will be divided into 2 categories:

1. Prelingual patients: subdivided into 3 groups

   * Cochlear implant recipient with no medical or radiological issues.
   * Cochlear implant recipients with medical concern or with other disabilities as syndromic patients.
   * Cochlear implant recipients with radiological issues.
2. Postlingual patients: subdivided into 3 groups

   * Cochlear implant recipients with no medical or radiological issues.
   * Cochlear implant recipients with medical concern or with other disabilities as syndromic patients.
   * Cochlear implant recipients with radiological issues.

Inclusion criteria:

Patients who received cochlear implant at Sohag university hospital and fulfill the following criteria:

* Age: from one year up to 60.
* Prelingual who had one year of regular speech therapy
* Postlingual patients.

  • Method:
  1. Background information:

     * History: Age, gender, Age at which hearing loss occur, cause of hearing loss, duration of hearing loss.
     * Family support.
     * Expectation of patient (if post lingual patient).
     * Expectation of parents.
  2. Hearing assessment:
* Aided Pure Tone Audiometry (PTA) level.
* Speech perception

  1. speech perception threshold (SRT).
  2. Speech perception in quiet for patients who developed language and postlingual patients using phonetically Balanced words for kinder garden ( PBKG) words, phonetically balanced words for adult (PBA), word intelligibility by picture identification (WIPI) or minimal birds.
  3. Speech in noise test: for patients who developed language and post lingual patients.

     3- Impedance telemetry. 4- Electrically evoked action potential (ECAP). 5- Cortical evoked P1N1 potential. Informed written consent will be taken from all Participant patients or their legal guardians.

     This search will submit for approval from Research Ethics committee of Sohag Faculty of medicine.

     All investigation will be done cost free.

ELIGIBILITY:
Inclusion Criteria:

-

Patients who received cochlear implant at Sohag university hospital and fulfill the following criteria:

* Age: from one year up to 60.
* Prelingual who had one year of regular speech therapy
* Postlingual patients.

Exclusion Criteria:

* none

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cochlear implant recipients in Sohag University Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Hearing threshold for Cochlear implant users at Sohag University Hospital | one year postoperative
  Pure Tone Audiometery will be used to measure the hearing threshold in decible at each frequnecy from 250 Hz to 8000 Hz
Central processing of speech for cochlear implant users at Sohag university Hospital | one year postoperative
  Auditory Evoked Potential for detection of P1 wave which generated at central auditory area, Presence of P1 wave means normal speech processing, while absence of P1 wave means abnormal speech processing

CONTACTS AND LOCATIONS:
Overall Officials: Shahenda A Moussa, Master, Principal Investigator — Sohag university, Faculty of medicine

IPD SHARING:
Plan to Share IPD: No
undecided

REFERENCES:
- [Background] Korver AM, Smith RJ, Van Camp G, Schleiss MR, Bitner-Glindzicz MA, Lustig LR, Usami SI, Boudewyns AN. Congenital hearing loss. Nat Rev Dis Primers. 2017 Jan 12;3:16094. doi: 10.1038/nrdp.2016.94. PMID 28079113